CLINICAL TRIAL: NCT06275269
Title: Comparison of the Safety and Economics of Translaryngeal Endoscopic Mucosal Injection Versus Ultrasound-Guided Injection of Triamcinolone for the Treatment of Subglottic Stenosis: a Multicenter, Randomized Controlled Study.
Brief Title: Endoscopic Mucosal Injection Versus Ultrasound-Guided Injection of Triamcinolone to Treat Subglottic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZRJY2021-BJ08-04-02
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Subglottic Stenosis
Keywords: Subglottic Stenosis; Triamcinolone; Translaryngeal Endoscopic Mucosal Injection; Ultrasound-Guided Injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-Guided Triamcinolone Injection Treatment Group (Experimental): Ultrasound-Guided Triamcinolone Injection for the Treatment of Subglottic Stenosis
  Interventions: Procedure: Ultrasound-Guided
- Translaryngeal Endoscopic Mucosal Injection of Triamcinolone Treatment Group (Experimental): Translaryngeal Endoscopic Mucosal Injection for the Treatment of Subglottic Stenosis
  Interventions: Procedure: Translaryngeal Endoscopic Mucosal Injection

INTERVENTIONS:
Procedure: Ultrasound-Guided — Ultrasound-Guided Triamcinolone Injection
  Arms: Ultrasound-Guided Triamcinolone Injection Treatment Group
Procedure: Translaryngeal Endoscopic Mucosal Injection — Translaryngeal Endoscopic Mucosal Injection of Triamcinolone
  Arms: Translaryngeal Endoscopic Mucosal Injection of Triamcinolone Treatment Group

SUMMARY:
This study employs a multicenter, randomized controlled trial method, where patients meeting the inclusion criteria for subglottic stenosis are randomly divided into two groups. These groups are respectively undergoing translaryngeal endoscopic mucosal injection and ultrasound-guided injection of triamcinolone treatment. The comparison will focus on various indicators such as therapeutic effect, incidence of adverse reactions, treatment costs, and hospital resource utilization between the two groups. The safety and effectiveness will be compared to determine the relative merits of the two treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* 1: "Diagnosed with subglottic stenosis through laryngoscopic examination or imaging studies such as CT."
* 2: "Experiencing symptoms related to subglottic stenosis, such as breathing difficulties, hoarseness, etc."

Exclusion Criteria:

* 1: "Severe cardiopulmonary dysfunction, patients extremely debilitated and unable to tolerate the procedure."
* 2: "Patients allergic to lidocaine, midazolam, triamcinolone, or any of their components."
* 3: "Pregnant or lactating women."
* 4: "Unstable angina, congestive heart failure, severe bronchial asthma."
* 5: "Severe hypertension and arrhythmias, hemodynamically unstable, and severe respiratory failure (PaO2 <60mmHg after oxygen therapy or mechanical ventilation)."
* 6: "Known coagulation dysfunction, inability to stop anticoagulants, antiplatelet agents, aspirin, or nonsteroidal anti-inflammatory drugs before treatment."
* 7: "Patients do not agree to participate in this study."
* 8: "Participation in other studies within the last three months and not withdrawn or concluded, or having received triamcinolone treatment less than 1 month ago."
* 9: "Researchers believe there are any circumstances making the patient unsuitable for inclusion."

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Short-Term Postoperative Complications | one week after intervention
  Follow-up on short-term postoperative complications (including pneumothorax, bleeding, wound infection, pain, fever, etc.)

SECONDARY OUTCOMES:
Overall medical expenses incurred by patients | one week after intervention
  Overall medical expenses incurred

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No